CLINICAL TRIAL: NCT01927718
Title: A Pilot Study of Thalidomide to Overcome Lenalidomide Resistance in Patients Suffering Biochemical Progression on Maintenance Therapy After Autologous Hematopoietic Stem Cell Transplantation for Multiple Myeloma
Brief Title: Thalidomide to Overcome Lenalidomide Resistance After Autologous Hematopoietic Stem Cell Transplantation (HCT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Response Rate
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0806; NCI-2014-00157 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Myeloma
Keywords: Blood And Marrow Transplantation; Myeloma; Multiple myeloma; MM; Autologous stem cell transplantation; ASCT; Thalidomide; Thalomid; Lenalidomide; CC-5013; Revlimid; Questionnaires; Surveys
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Thalidomide; Lenalidomide; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide + Lenalidomide (Experimental): Thalidomide 100 mg by mouth daily for 28 days in a 28 day cycle started after the clinical documentation of biochemical progression.
  Lenalidomide continued by mouth at the previous dose of 5 mg daily for 21 days on a 28 day cycle, 5 mg daily for 28 days on a 28 day cycle, 10 mg daily for 28 days on a 28 day cycle, or 15 mg daily for 28 days on a 28 day cycle.
  Interventions: Drug: Thalidomide; Drug: Lenalidomide; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Thalidomide — 100 mg by mouth daily for 28 days in a 28 day cycle.
  Other Names: Thalomid
Drug: Lenalidomide — Lenalidomide continued by mouth at the previous dose of 5 mg daily for 21 days on a 28 day cycle, 5 mg daily for 28 days on a 28 day cycle, 10 mg daily for 28 days on a 28 day cycle, or 15 mg daily for 28 days on a 28 day cycle.
  Other Names: CC-5013; Revlimid
Behavioral: Questionnaires — Questionnaire completion at screening, once a month for the first 6 months, then every other month while on study.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if adding low dose Thalidomide (thalidomide) to Revlimid (lenalidomide) maintenance therapy will help control MM after an autologous stem cell transplant. Researchers also want to learn if treatment with these study drugs will improve participants' quality of life.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will begin taking lenalidomide and thalidomide by mouth once a day, in the evening. Thalidomide should be taken at least 1 hour after your evening meal. Bedtime is the best time to take thalidomide.

Swallow the lenalidomide and thalidomide capsules whole with at least 4 ounces of water. Do not open, crush, or break the lenalidomide or thalidomide capsules. If you touch a broken lenalidomide or thalidomide capsule, wash the affected area of your body with soap and water.

If you miss a dose of lenalidomide and/or thalidomide, and it has been less than 12 hours since your regular dosing time, take it as soon as you remember. If it has been more than 12 hours, just skip your missed dose. Do not take 2 doses at the same time.

If you take too much lenalidomide and/or thalidomide (overdose), call your primary healthcare provider or poison control center right away.

If you vomit after taking your dose, you should wait to take another dose until the next scheduled time.

You will be given a patient study drug diary. You will use this diary to write down what time you took each dose of lenalidomide and thalidomide. You need to bring the study drug diary to every study visit so the study staff can review it.

Since lenalidomide and thalidomide both increase the risk of developing blood clots, especially in patients who are at high risk or with a history of blood clots, you may receive heparin, warfarin, or aspirin to help prevent blood clots. Your doctor will decide which medication you need, or your doctor may decide that you do not need a medication to help prevent blood clots, based on your platelet count (cells that help your blood clot).

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Visits:

Once a month for the first 6 months:

* You will have a physical exam.
* You will have a neurological exam (tests to check the functioning of your nerves, including tests of your balance and reflexes). You will be asked about any numbness or tingling you may be experiencing.
* Blood (about 2 tablespoons) and urine will be collected for routine tests, liver and kidney function tests, blood clotting tests (if needed), and tests to check the status of the disease.

If the doctor thinks the disease has either gone into remission (gotten better) or has gotten worse, you will have additional blood tests and a bone marrow biopsy to check the status of the disease.

After Month 6, during every even-numbered month you are on study (Months 8, 10, 12, and so on), blood (about 2 tablespoons) and urine will be collected for routine tests and to check the status of the disease.

Questionnaires:

You will be asked to complete a questionnaire about your symptoms and quality of life during screening, once a month for the first 6 months, and then every other month while you are on study.

You will sometimes fill out the questionnaire by hand on a piece of paper, or you may be asked the questions over the telephone by a member of the study staff. Other times, the questionnaire will be done over the phone with an automated phone system. The telephone system will ask you to rate how strong and tolerable the symptoms are, and how much the symptoms interfere with your daily life. Rating your symptoms using the telephone system should take less than 5 minutes for each call. The research nurse will teach you how to use the automated telephone system.

Length of Treatment:

You will receive the study drugs for up to 2 years. You will no longer be able to take the study drug if the doctor thinks it is in your best interest, if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions or keep appointments.

Your participation on the study will be over after the end-of-study visit.

End-of-Study Visit:

About 30 days of your last dose of study drugs:

* You will have a physical exam and neurological exam.
* Blood (about 2 tablespoons) and urine will be collected for routine tests and to check the status of the disease.
* You will have a bone marrow biopsy to check the status of the disease, if your doctor thinks it is needed.

This is an investigational study. Lenalidomide and Thalidomide are FDA approved and commercially available for the treatment of myeloma. The use of these chemotherapy drugs in treating MM that has gotten worse after treatment with lenalidomide is considered investigational. The study doctor can explain how the study drug(s) are designed to work.

Up to 17 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative able to sign an informed consent form.
2. Age 18 years old or older.
3. Multiple myeloma showing signs of biochemical progression while taking lenalidomide or lenalidomide plus dexamethasone maintenance therapy after autologous hematopoietic stem cell transplantation. (Progression is defined solely based on serum or urine M-protein, or in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved serum free light chain level -- please also see appendix E for full details.)
4. Patients with biochemical progression only with at least >/= 25% increase from the baseline in any of the following parameters on at least 2 occasions; and when the treating physician deems a change in therapy is necessary: a. Serum M-protein; b. Urine M-protein; or, c. In patients without measureable serum and urine M-protein levels; the difference between involved and uninvolved free light chain levels.
5. Lenalidomide must have been used for at least 6 months after autologous hematopoietic stem cell transplantation with the current dose of Lenalidomide 15 mg/day or less.
6. Serum creatinine clearance (Cockcroft-Gault Equation) >= 50 mL/minute.
7. Performance score of at least 80% by Karnofsky or 0 to 2 Eastern Cooperative Oncology Group (ECOG).
8. Patients must be informed of the Celgene Risk Management Program and mandatory registration as well as be willing and able to comply with its requirements.
9. Negative Beta Human Chorionic Gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization and willing to ongoing pregnancy testing while on treatment with lenalidomide.
10. Woman with child bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME.
11. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
12. Laboratory test results within these ranges: a. Absolute neutrophil count > 1000 cells/mm3. b. Platelet count > 50,000 cells/mm3 for patients with < 50% of bone marrow plasma cells OR platelet count > 25,000 cells/mm3 for patients in whom > 50% of the bone marrow nucleated cells were plasma cells. c. Total bilirubin </= 2.0 mg/dL. d. AST (SGOT) and ALT (AGPT) </= 3 x upper normal limit.
13. Able to take anticoagulation, warfarin or equivalent agent, as detailed in the treatment plan.
14. HIV negative.

Exclusion Criteria:

1. Any serious medical condition or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Patients with symptomatic relapse, including those with new bone lesions, soft tissue plasmacytomas, an increase in the size of existing bone lesions or soft tissue plasmacytomas, decrease in hemoglobin, rise in serum creatinine or hypercalcemia.
3. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
4. Known hypersensitivity to thalidomide or lenalidomide.
5. Known history of resistance to Thalidomide.
6. Patients with grade III-IV neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Bashir, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2014 to august 2016. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Thalidomide + Lenalidomide: Thalidomide 100 mg by mouth daily for 28 days; Lenalidomide continued by mouth at the previous dose of 5 mg daily for 21 days on a 28 day cycle, 5 mg daily for 28 days on a 28 day cycle, 10 mg daily for 28 days on a 28 day cycle, or 15 mg daily for 28 day cycle.
Period: Overall Study
Arm/Group | Thalidomide + Lenalidomide
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Thalidomide + Lenalidomide: Thalidomide 100 mg by mouth daily for 28 days and Lenalidomide continued by mouth at the previous dose of 5 mg daily for 21 days on a 28 day cycle, 5 mg daily for 28 days on a 28 day cycle, 10 mg daily for 28 days on a 28 day cycle, or 15 mg daily for 28 day cycle.
Arm/Group | Thalidomide + Lenalidomide
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Primary endpoint is response rate (RR) measured by the proportion of patients receiving the combination, whose disease stabilizes, or returns to at least its previous response level prior to progression, assessed at 3-months after starting the combination.1.Stringent Complete Remission (sCR): Follows criteria for CR, plus:Normal FLC ratio, Absence of clonal cells in the BM; Complete Remission (CR) All of the following criteria are met:Negative SIFE and UIFE:Disappearance of any soft tissue plasmacytomas:< 5% plasma cells in the BM. 2.Very Good Partial Response (VGPR):One or more of the following must be present:Serum and urine M-protein detectable by immunofixation but not on electrophoresis:≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours.Partial Response (PR) Both of the following must be present:≥ 50% reduction in SPEP:Reduction in 24-hour UPEP by ≥ 90% or to < 200 mg/24 hours.3.Stable Disease (SD)Does not meet the criteria for CR, VGPR, PR, or PD.4.Pr
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Thalidomide + Lenalidomide
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse event collection with 28 day treatment cycle, and up to 30 days after the last dose of the study drugs.
Arm/Group | Thalidomide + Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide + Lenalidomide (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Elevated alanine transaminase (ALT) (Investigations) | 1 (1)
Elevated Aspartate aminotransferase (AST) (Investigations) | 1 (1)
Elevated creatinine (Investigations) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Infection (Investigations) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2)
Loss of balance (Investigations) | 1 (1)
Low white blood count (Investigations) | 2 (2)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nerve pain (Nervous system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
paraesthesia (Nervous system disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes